CLINICAL TRIAL: NCT03692182
Title: Antipsychotic Use Within the Program of All-inclusive Care for the Elderly (PACE)
Brief Title: The Use of Antipsychotics in the Program of All-inclusive Care for the Elderly (PACE)
Status: Completed | Type: Observational
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: AP-BPSD-001
Record Dates: First submitted 2018-09-25; First posted 2018-10-02 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Behavioral and Psychiatric Symptoms of Dementia
Keywords: Antipsychotic; Dementia
MeSH Terms: conditions — Behavior; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Participants enrolled in PACE who received an antipsychotic medication.

SUMMARY:
The aim of this study is to retrospectively evaluate and describe the use of antipsychotics among participants enrolled in the Program of All-inclusive Care for the Elderly (PACE), a community-based practice setting.

DETAILED DESCRIPTION:
Much national attention has been given to assessing and reducing the use of antipsychotics among nursing home residents, yet comparatively little attention has focused on antipsychotic use among older adults receiving care in community-based settings. The primary objective of this study is to determine the prevalence of antipsychotic use among a nationally representative sample of nursing home-eligible older adults in a community-based practice setting known as Program of All-inclusive Care for the Elderly (PACE). The secondary objectives are focused on characterizing antipsychotic use within PACE and for these participants. Specifically, the investigator's secondary objectives are to describe patterns of other drugs concomitantly used with antipsychotics (e.g., benzodiazepines, opioids) and to identify clinically relevant drug-drug interactions involving antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Participant enrolled in PACE contractually receiving pharmacy services from Tabula Rasa Healthcare CareKinesis Pharmacy (Tabula Rasa HealthCare) during the project time period (January 2017 through December 2017).

Exclusion Criteria:

* Participant with a diagnosis of bipolar disorder and/or schizophrenia, according to pharmacy records.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Program of All-inclusive Care for the Elderly (PACE) is a Medicare-Medicaid program that provides comprehensive medical and supportive services to individuals >55 years of age who are certified by their state as needing nursing home care but are able to live safely in the community through PACE, as an alternative to institutionalization.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Antipsychotic Use | 12 months
  Quantitative description of antipsychotic use as assessed by pharmacy records

SECONDARY OUTCOMES:
Concomitant Drug Use with Antipsychotics | 12 months
  Qualitative and quantitative description of patterns of other drugs concomitantly used with antipsychotics as assessed by pharmacy records
Drug-Drug Interactions | 12 months
  Qualitative and quantitative description of drug-drug interactions involving antipsychotics as assessed by proprietary clinical decision support system (CDSS)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin T Bain, PharmD, MPH, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare, Moorestown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There will be no disclosure of participant information and no details of participant identity will be part of any presentation or publication of the research. Participant confidentiality will be held in strict trust by the project investigators. The project data or other information generated will be held in strict confidence. No information concerning the project or the data will be released to any unauthorized third party without prior written consent.

REFERENCES:
- [Background] Bain KT, Schwartz EJ, Chan-Ting R. Reducing Off-Label Antipsychotic Use in Older Community-Dwelling Adults With Dementia: A Narrative Review. J Am Osteopath Assoc. 2017 Jul 1;117(7):441-450. doi: 10.7556/jaoa.2017.090. PMID 28662557
- [Background] Pimentel CB, Donovan JL, Field TS, Gurwitz JH, Harrold LR, Kanaan AO, Lemay CA, Mazor KM, Tjia J, Briesacher BA. Use of atypical antipsychotics in nursing homes and pharmaceutical marketing. J Am Geriatr Soc. 2015 Feb;63(2):297-301. doi: 10.1111/jgs.13180. PMID 25688605
- [Background] Liperoti R, Pedone C, Corsonello A. Antipsychotics for the treatment of behavioral and psychological symptoms of dementia (BPSD). Curr Neuropharmacol. 2008 Jun;6(2):117-24. doi: 10.2174/157015908784533860. PMID 19305792
- [Background] Schneider LS, Dagerman KS, Insel P. Risk of death with atypical antipsychotic drug treatment for dementia: meta-analysis of randomized placebo-controlled trials. JAMA. 2005 Oct 19;294(15):1934-43. doi: 10.1001/jama.294.15.1934. PMID 16234500
- [Background] Salvo F, Pariente A, Shakir S, Robinson P, Arnaud M, Thomas S, Raschi E, Fourrier-Reglat A, Moore N, Sturkenboom M, Hazell On Behalf Of Investigators Of The Aritmo Consortium L; Investigators of the ARITMO Consortium. Sudden cardiac and sudden unexpected death related to antipsychotics: A meta-analysis of observational studies. Clin Pharmacol Ther. 2016 Mar;99(3):306-14. doi: 10.1002/cpt.250. Epub 2015 Nov 20. PMID 26272741
- [Background] Gareri P, De Fazio P, Manfredi VG, De Sarro G. Use and safety of antipsychotics in behavioral disorders in elderly people with dementia. J Clin Psychopharmacol. 2014 Feb;34(1):109-23. doi: 10.1097/JCP.0b013e3182a6096e. PMID 24158020
- [Background] Mehta S, Johnson ML, Chen H, Aparasu RR. Risk of cerebrovascular adverse events in older adults using antipsychotic agents: a propensity-matched retrospective cohort study. J Clin Psychiatry. 2010 Jun;71(6):689-98. doi: 10.4088/JCP.09m05817yel. PMID 20573328